CLINICAL TRIAL: NCT04680130
Title: Clinico-Pathologic-Genetic-Imaging Study of Neurodegenerative and Related Disorders
Acronym: AND1
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Keith A. Josephs, Professor of Neurology, Mayo Clinic
Other Study IDs: 19-009999
Record Dates: First submitted 2020-11-03; First posted 2020-12-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: PSP; CBD; PCA; LPA; Semantic Dementia; Semantic Aphasia; Behavioral Variant of Frontotemporal Dementia; FTD; PPA; Apraxia of Speech; MSA - Multiple System Atrophy; Parkinson Disease
MeSH Terms: conditions — Frontotemporal Dementia; Aphasia; Pick Disease of the Brain; Apraxias; Shy-Drager Syndrome; Parkinson Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurodegenerative symptoms
  Interventions: Drug: C-11 PiB; Drug: AV1451 Tau; Drug: C-11 ER176

INTERVENTIONS:
Drug: C-11 PiB — Completing PET scan looking for amyloid protein
Drug: AV1451 Tau — Completing PET scan looking for tau protein
Drug: C-11 ER176 — Completing PET scan looking for neuroinflammation

SUMMARY:
The investigators aim to learn more about symptoms suggestive of a neurodegenerative process.

DETAILED DESCRIPTION:
The investigators will recruit participants with symptoms suggestive of a neurodegenerative and/or related disease. Participants could be evaluated on a yearly basis, undergoing a baseline visit and possible follow-up evaluations with an interval of one year. At each visit, participants could undergo any combination of the following based on their symptoms and complaints: a neurological assessment, a speech/language assessment, a neuropsychometric assessment, an MRI, an FDG PET/CT scan, a PiB PET/CT scan, a Tau PET/CT scan and/or a C-11 ER176 PET/CT scan. All participants will be asked to provide a blood sample to allow for future genetic studies.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be over the age of 21
* Have symptoms suggestive of a neurodegenerative and/or related disorder

Exclusion Criteria:

* Participants will be excluded if they have any concurrent illnesses that could account for all of their symptoms, such as traumatic brain injury, encephalitis, strokes or developmental syndromes
* Women that are pregnant or post-partum and breast-feeding will be excluded
* Participants will be excluded if they have any of the following genetic conditions which can increase the chance of cancer: Cowden disease, Lynch syndrome, Hypogammaglobulinemia, Wiskott-Aldrich syndrome and Down's syndrome
* Participants will be excluded if MRI is contraindicated (metal in head, cardiac pace maker, etc), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma, intracranial neoplasm or large cortical infarcts)
* Participants will be excluded if they are medically unstable or are on medications that might affect brain structure or metabolism (e.g. chemotherapy)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptoms of neurodegenerative disease
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2050-11 (Estimated); Study Completion 2050-11 (Estimated)

PRIMARY OUTCOMES:
Imaging analysis | 1 year
  Longitudinal images and correlates will be measured and tracked to determine direct correlations in the brain with disease progression on a yearly basis

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials